CLINICAL TRIAL: NCT06546553
Title: FIRST-IN-HUMAN (FIH), OPEN-LABEL, PHASE 1 DOSE ESCALATION AND EXPANSION STUDY DESIGNED TO EVALUATE THE SAFETY, TOLERABILITY, PK, PD, AND PRELIMINARY CLINICAL ACTIVITY OF PF-07826390 AS A SINGLE AGENT OR IN COMBINATION TREATMENT FOR PARTICIPANTS WITH ADVANCED SOLID TUMORS.
Brief Title: A Study to Learn About How Different Amounts of the Study Medicine PF-07826390 Act in the Body of People With Cancer When Taken Alone or With Other Anti-cancer Medicines.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated as part of strategic considerations and not based on safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C5321001; NCT06546553 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-07-22; First posted 2024-08-09 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Neoplasms; Non-small-cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck; Renal Cell Carcinoma; Colorectal Carcinoma; Ovarian Carcinoma
Keywords: Solid tumors; metastatic; advanced; micro satellite stable; anti-PD-1; PF-07282690; LILRB12; sasanlimab; PD-1 resistance; PD-1 naive; PDx resistance; PDxnaive; Carcinoma, Non-Small Cell Lung; Non-Small Cell Lung Cancer; Non-Small Cell Lung Carcinoma; Non-Small-Cell Lung Carcinoma; Nonsmall Cell Lung Cancer; Colorectal Cancer; Colorectal Neoplasms; Colorectal Carcinoma; Colorectal Tumors; Renal Cell Carcinoma; Kidney Neoplasms; Rectal Disease; Neoplasms, Colorectal; Malignant Melanoma; Microsatellite Stable Colorectal Cancer (MSS CRC)
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Colorectal Neoplasms; Ovarian Neoplasms; Neoplasm Metastasis; Kidney Neoplasms; Rectal Diseases; Melanoma | interventions — Leukocyte Immunoglobulin-like Receptor B1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1A: PF-07826390 Monotherapy (Experimental): PF-07826390 monotherapy at prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07826390
- Part 1B: PF-07826390 + sasanlimab (Experimental): PF-07826390 + sasanlimab at prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07826390; Biological: sasanlimab
- Part 2A (Arm 1): PF-07826390 + sasanlimab (Experimental): PF-07826390 + sasanlimab dose expansion in NSCLC 2L+ at prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07826390; Biological: sasanlimab
- Part 2A (Arm 2): PF-07826390 + sasanlimab (Experimental): PF-07826390 + sasanlimab dose expansion in MSS CRC 2L+ at prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07826390; Biological: sasanlimab
- Part 2A (Arm 3): PF-07826390 + sasanlimab (Experimental): PF-07826390 + sasanlimab dose expansion in RCC 2L+ at prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07826390; Biological: sasanlimab
- Part 2B: PF-07826390 (Experimental): PF-07826390 dose expansion in NSCLC 2L+ at prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07826390
- Part 2C: PF-07826390 + SOC (Experimental): PF-07826390 + SOC (anti-PD-1 + platinum -based chemo) dose expansion for a PDx-naive NSCLC 1L at prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07826390; Other: SOC (anti-PD-1 + platinum -based chemo)

INTERVENTIONS:
Drug: PF-07826390 — PF-07826390 is a novel, fully humanized bispecific IgG1 that targets the leukocyte immunoglobulin-like receptor, LILRB1 and LILRB2 (B1 and B2) cell-surface receptors
  Other Names: LILRB1/2
Biological: sasanlimab — A monoclonal antibody that blocks the interaction between PD-1 and PD-L1/L2
  Other Names: PF-06801591
  Arms: Part 1B: PF-07826390 + sasanlimab; Part 2A (Arm 1): PF-07826390 + sasanlimab; Part 2A (Arm 2): PF-07826390 + sasanlimab; Part 2A (Arm 3): PF-07826390 + sasanlimab
Other: SOC (anti-PD-1 + platinum -based chemo) — Standard of Care (anti-PD-1 + platinum -based chemo)
  Arms: Part 2C: PF-07826390 + SOC

SUMMARY:
The purpose of this study is to learn about the:

* safety (the effect of the study medicine on the participant's body),
* effects of the study medicine alone or in combination with sasanlimab -
* the best amount of the study medicine.

This study is seeking participants who have solid tumors (An abnormal mass of tissue) that:

* have advanced (cancer that does not disappear or stay away with treatment) or
* are metastatic (has spread to other parts of the body).

This includes (but limited to) the following cancer types:

* Non-Small Cell Lung Cancer (NSCLC): It's a type of lung cancer where the cells grow slowly but often spread to other parts of the body.
* Colorectal Cancer (CRC): This is a disease where cells in the colon or rectum grow out of control.
* Renal Cell Carcinoma (RCC): This is a cancer that starts in the kidney.

All participants in this study will receive the study medication (PF-07826390) as an IV infusion (given directly into a vein) at the study once every four weeks in 28 day cycles.

The study participants depending on the group enrolled in, will receive the study medication (PF-07826390 alone or in combination with other anti-cancer medications (sasanlimab). Sasanlimab is given as a shot under the skin every 4 weeks.

Participants can continue to take the study medication (PF-07826390) until their cancer is no longer responding. Participants who are taking sasanlimab may receive it for up to 2 years.

The study will look at the experiences of people receiving the study medicines. This will help see if the study medicines are safe and effective.

Participants will be involved in this study for up to 4 years. During this time, participants will have a study visit every week. The participants after stopping the study medicine (at about 2 years) will be followed for another two years to see how the participants are doing.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of advanced, unresectable, and/or metastatic or relapsed/refractory solid tumor
* Part 1A: Participants with solid tumors where anti-PD-(L)1 is an established treatment. Participants must have progressed on or following prior anti-PD-(L)1 therapy if approved, available, tolerable, and eligible
* Part 1B: Participants either meeting Part 1A criterion, or participants with "cold" solid tumors where anti-PD-(L)1 therapy is not an established treatment
* Part 2: Participants with NSCLC (2A Arm 1 and 2B) must have received platinum-based chemotherapy and anti-PD-(L)1 or have intolerability to or refusal of standard therapies. Participants with NSCLC who have not been previously treated with a prior anti-pd-(L) will be enrolled in Part 2C.
* Participants with MSS CRC (Part 2A Arm 2) must have received fluoropyrimidine-, oxaliplatin, and irinotecan-based chemotherapy, an anti-VEGF agent and anti-EGFR inhibitor (if RAS wildtype) and/or other molecularly targeted therapy if appropriate. Participants with RCC (Part 2A Arm 3) must have received prior tyrosine kinase inhibitor (TKI), anti-PD-(L)1 (if not receiving anti-PD-1 on protocol), anti-CTLA-4 (optional), hypoxia-inducible factor 2 alpha (HIF2a) inhibitor, or mTOR inhibitor or have documented intolerance to the standard therapy.
* At least 1 measurable lesion based on RECIST 1.1 that has not been previously irradiated (Part 1 exceptions permitted after review and approval)
* Able to provide pre-treatment (and optional on-treatment) tumor tissue

Exclusion Criteria:

* Treatment with any systemic anticancer therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to planned first dose
* Active or history of clinically significant autoimmune disease or other medical condition that required chronic systemic immunosuppressive therapy within recent 2 years
* Prior treatment with another LILRB1 (ILT2), LILRB2 (ILT4), and/or LILRB1/2 (B1 and B2) antagonist antibodies or pathway targeting agents, including HLA conformers and HLA-G antibodies.
* Lack of adequate organ (bone marrow, renal, liver) function
* History of severe immune-mediated adverse event or cytokine release syndrome that was considered related to prior immune modulatory therapy that required immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
PART 1: Number of participants with Dose-limiting toxicities (DLT) | First cycle, Day 1 up to Day 28
  Any of the prespecified AEs that are attributable to one, the other, or both study treatments, occurring in the DLT observation period are considered DLTs, excluding toxicities clearly due to underlying disease or extraneous causes.
PART 1 & 2: Incidence of Adverse Events (AE)s | From start of the treatment and up to 90 days after last dose or start of new anticancer therapy, whichever occurred first.
  An adverse event (AE) is any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it. SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/ incapacity; congenital anomaly. AEs included both serious and all non-serious AEs.
PART 1 & 2: Number of participants with laboratory abnormalities | From start of the treatment and up to 90 days after last dose or start of new anticancer therapy, whichever occurred first.
  Number of participants with laboratory test abnormalities. Laboratory test parameters included hematology, coagulation, liver function, renal function, electrolytes, clinical chemistry, and urinalysis (dipstick and microscopy).
Part 2: Objective Response - Number of Participants With Objective Response | Baseline and every 8 to 12 weeks through time of confirmed disease progression, death, unacceptable toxicity, or through study completion, approximately 2 years.
  Percentage of participants with objective response-based assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by the Investigator.

SECONDARY OUTCOMES:
Objective Response - Number of Participants with Objective Response | Baseline and every 8 to 12 weeks through time of confirmed disease progression, death, unacceptable toxicity, or through study completion, approximately 2 years
  Percentage of participants with objective response-based assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by the Investigator
Time to event endpoints: duration of response (DOR) by RECIST v1.1 | Baseline to confirmed disease progression, up to 2 years after the last dose of study treatment
  Time to event: DOR according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) as assessed by the Investigator.
Time to event endpoints: progression-free survival (PFS) by RECIST v1.1 | Baseline to confirmed disease progression, up to 2 years after the last dose of study treatment
  Time to event: PFS according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) as assessed by the Investigator.
Part 1: Maximum Observed Serum Concentration (Cmax) | Cycle 1 Day 1, 2, 3, 8, 15 and 22; Cycle 2 Day 1 and 15; Cycle 3+ Day 1 (each cycle is 28 days)
  Cycle 1: Pre-dose, 1, 4, 8, 24, 48, 168, 336 and 504 hours post dose. Cycle 2: Pre-dose and 336 hours post dose. Cycle 3: Pre-dose, 1, 4, 24, 168 and 336 hours post dose. Cycle 3 and beyond Pre-dose only.
Part 1: Time to Reach Maximum Serum Concentration (Tmax) of PF-07826390 | Cycle 1 Day 1, 2, 3, 8, 15 and 22; Cycle 2 Day 1 and 15; Cycle 3+ Day 1 (each cycle is 28 days)
  Cycle 1: Pre-dose, 1, 4, 8, 24, 48, 168, 336 and 504 hours post dose. Cycle 2: Pre-dose and 336 hours post dose. Cycle 3: Pre-dose, 1, 4, 24, 168 and 336 hours post dose. Cycle 3 and beyond Pre-dose only.
Part 1: Serum Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-07826390 | Cycle 1 Day 1, 2, 3, 8, 15 and 22; Cycle 2 Day 1 and 15; Cycle 3+ Day 1 (each cycle is 28 days)
  Cycle 1: Pre-dose, 1, 4, 8, 24, 48, 168, 336 and 504 hours post dose. Cycle 2: Pre-dose and 336 hours post dose. Cycle 3: Pre-dose, 1, 4, 24, 168 and 336 hours post dose. Cycle 3 and beyond Pre-dose only.
Part 1: Serum Area Under the Curve From Time Zero to Last Time Zero to clearance (CL/F) of PF-07826390 | Cycle 1 Day 1, 2, 3, 8, 15 and 22; Cycle 2 Day 1 and 15; Cycle 3+ Day 1 (each cycle is 28 days)
  Cycle 1: Pre-dose, 1, 4, 8, 24, 48, 168, 336 and 504 hours post dose. Cycle 2: Pre-dose and 336 hours post dose. Cycle 3: Pre-dose, 1, 4, 24, 168 and 336 hours post dose. Cycle 3 and beyond Pre-dose only.
Part 1: Serum under the curve apparent volume of distribution during terminal phase (Vz/F) of PF-07826390 | Cycle 1 Day 1, 2, 3, 8, 15 and 22; Cycle 2 Day 1 and 15; Cycle 3+ Day 1 (each cycle is 28 days)
  Cycle 1: Pre-dose, 1, 4, 8, 24, 48, 168, 336 and 504 hours post dose. Cycle 2: Pre-dose and 336 hours post dose. Cycle 3: Pre-dose, 1, 4, 24, 168 and 336 hours post dose. Cycle 3 and beyond Pre-dose only.
Part 1: Serum under the curve terminal elimination half life (T ½) of PF-07826390 | Cycle 1 Day 1, 2, 3, 8, 15 and 22; Cycle 2 Day 1 and 15; Cycle 3+ Day 1 (each cycle is 28 days)
  Cycle 1: Pre-dose, 1, 4, 8, 24, 48, 168, 336 and 504 hours post dose. Cycle 2: Pre-dose and 336 hours post dose. Cycle 3: Pre-dose, 1, 4, 24, 168 and 336 hours post dose. Cycle 3 and beyond Pre-dose only.
Part 1 and Part 2: Serum Concentrations of PF-07826390 in combination (Part 1B, 2A and 2C) | Prior to dosing at Cycle 1+ Day 1 until last dose of study treatment, approximately 2 years (each cycle is 28 days)
  Day 1 (all cycles) and EOT.
Part 1 and Part 2: Incidence and titers of antidrug antibodies (ADA) against PF-07826390 | Prior to dosing at Cycle 1+ Day 1 up to end of study treatment, approximately 2 years (each cycle is 28 days)
  Day 1 (all cycles) and end of treatment
Part 1 and Part 2: Paried Tumor Biopsies | Baseline through Cycle 2 Day 15 (each cycle is 28 days)
  Pre-dose and C2 Day 15
Part 2: Time to Reach Maximum Serum Concentration (Tmax) of PF-07826390 | Cycle 1 Day 1 until last dose of study treatment, approximately 2 years (each cycle is 28 days)
  Cycle 1, 2 and 3: Pre-dose, 1, 24, and 336 hours post dose. Cycle 4 and beyond Pre-dose only.
Part 2: Maximum Observed Serum Concentration (Cmax) of PF-07826390 | Cycle 1 Day 1 until last dose of study treatment, approximately 2 years (each cycle is 28 days)
  Cycle 1, 2 and 3: Pre-dose, 1, 24, and 336 hours post dose. Cycle 4 and beyond Pre-dose only.
Part 1: Pharmacodynamic blood samples: Receptor occupancy | Cycle 1 Day 1 until last dose of study treatment, approximately 2 years (each cycle is 28 days)
  Cycle 1: Pre-dose, 48, 168 and 336 hours post dose. Cycle 2: Pre-dose and 336 hours post dose. Cycle 3 and beyond pre-dose only.
Part 2: Pharmacodynamic blood samples Receptor Occupancy | Cycle 1 Day 1 until last dose of study treatment, approximately 2 years (each cycle is 28 days)
  Cycle 1: Pre-dose, 24 and 336 hours post dose, Cycle 2: Pre-dose, 24 and 336 hours post dose. Cycle 3 and beyond pre-dose only.
Part 2: Serum Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-07826390 | Cycle 1 Day 1 until last dose of study treatment, approximately 2 years (each cycle is 28 days)
  Cycle 1, Cycle 2 and Cycle 3: Pre-dose, 1, 24 and 336 hours post dose.
Part 2: Serum Area Under the Curve From Time Zero to clearance (CL/F) of PF-07826390 | Cycle 1 Day 1 until last dose of study treatment, approximately 2 years (each cycle is 28 days)
  Cycle 1, Cycle 2 and Cycle 3: Pre-dose, 1, 24 and 336 hours post dose.
Part 2: Serum under the curve apparent volume of distribution during terminal phase (Vz/F) of PF-07826390 | Cycle 1 Day 1 until last dose of study treatment, approximately 2 years (each cycle is 28 days)
  Cycle 1, Cycle 2 and Cycle 3: Pre-dose, 1, 24 and 336 hours post dose.
Part 2: Serum under the curve terminal elimination half life (T ½) of PF-07826390 | Cycle 1 Day 1 until last dose of study treatment, approximately 2 years (each cycle is 28 days)
  Cycle 1, Cycle 2 and Cycle 3: Pre-dose, 1, 24 and 336 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Florida Cancer Specialists, Orlando, Florida
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - START Midwest, Grand Rapids, Michigan
  - START San Antonio, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5321001